CLINICAL TRIAL: NCT05668520
Title: A Pilot Study of Nutritional Status in Patients With Huntington's Disease
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Aberdeen (Other)
Responsible Party: Principal Investigator, Zosia Miedzybrodzka, Professor, University of Aberdeen
Other Study IDs: 2-095-19
Record Dates: First submitted 2022-09-30; First posted 2022-12-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- weight stable: stage 2 and 3 as defined by the UHDRS Total Functional Capacity score will be recruited. Ten will have reported at least 5% weight loss in a 12-month period,
  Interventions: Diagnostic Test: Body composition using a hand-held body fat monitor • Resting Metabolic Rate (RMR) using a ventilated hood system
- weight loss: stage 2 and 3 as defined by the UHDRS Total Functional Capacity score will be recruited. Ten will have reported at least 5% weight loss in a 12-month period,
  Interventions: Diagnostic Test: Body composition using a hand-held body fat monitor • Resting Metabolic Rate (RMR) using a ventilated hood system

INTERVENTIONS:
Diagnostic Test: Body composition using a hand-held body fat monitor • Resting Metabolic Rate (RMR) using a ventilated hood system — Consent Paperwork
  * Nutritional assessment using MNA and MUST questionnaires
  * 24-hour dietary recall assessment Body weight, height, waist circumference, mid upper arm and calf circumference
  Other Names: Nutritional assessment

SUMMARY:
It is known that weight loss is a poor prognostic marker in HD, but it is not known which dietary interventions are optimal at different stages of the disease. Current guidelines for HD treatment are informed only by studies in people with other causes of weight loss. Our long term goal is to create the evidence base for improved nutritional management in HD. This study will pilot the tools to inform the development of clinical trials protocols. We want to know which measures can be used by patients manifesting obvious clinical features of HD, and which are most helpful in detecting clinically meaningful changes in nutrition status.

DETAILED DESCRIPTION:
Huntington's disease (HD) is a complex autosomal dominant disorder of (generally) adult onset. The clinical features of HD are cognitive decline, psychiatric disturbance, personality change and movement disorder. Although by EU definition a rare disease, better management and establishment of clinics for care of HD around the world have led to recognition of that the condition is much more common than previously considered.

Grampian has one of the longest established clinics for managing HD worldwide, and we now care for more than 150 people at different stages in HD, making us one of the largest five specialist clinics in the UK. Members of our team have led the production of European guidelines for HD management, and within this project, we have highlighted the importance of nutrition in HD. Weight loss is well documented as a clinical feature of all stages of Huntington's disease (HD). However, its metabolic basis is poorly understood and appetite has not been formally studied in patients with the condition. Furthermore, the composition of weight loss - muscle or fat has been little studied and modern nutrition assessment tools have not been applied in this cohort. It is known that weight loss is a poor prognostic marker in HD, but it is not known which dietary interventions are optimal at different stages of the disease. Current guidelines for HD treatment are informed only by studies in people with other causes of weight loss. The long term goal of this study is to create the evidence base for improved nutritional management in HD. This study will pilot the tools to inform the development of clinical trials protocols. The aim is to identify which measures can be used by patients manifesting obvious clinical features of HD, and which are most helpful in detecting clinically meaningful changes in nutrition status.

ELIGIBILITY:
Inclusion Criteria:

* stage 2 or 3 Huntington disease

Exclusion Criteria:

* unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: manifesting Huntington disease patients of North of Scotland Huntington's clinic
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
satisfactory completion of body composition | assessed at study visit for each participant
  measurement of body composition using hand-held body fat monitor
measurement of resting metabolic rate | assessed at study visit for each participant
  measurement of Resting Metabolic Rate (RMR) using a ventilated hood system
measurement of body weight | assessed at study visit for each participant
  body weight in kg
measurement of height | assessed at study visit for each participant
  height in metres
completion of measurement of waist, arm and calf circumference | assessed at study visit for each participant
  measurement of waist circumference, mid upper arm and calf circumference using a tape measure
nutritional assessment | assessed at study visit for each participant
  estimation of energy, protein, carbohydrate and fat intake using MNA and MUST questionnaires

SECONDARY OUTCOMES:
variability of measures to power future grant applications | at end of study
  Descriptive statistics of each measurement by group

CONTACTS AND LOCATIONS:
Locations (1):
- Zosia Miedzybrodzka, Aberdeen, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
de-identified data sharing would be considered on request but would require additional permissions